CLINICAL TRIAL: NCT01445132
Title: Adoptive Cell Therapy for B-Cell Malignancies After Allogeneic Hematopoietic Stem Cell Transplantation With Costimulated, Tumor-Derived Lymphocytes
Brief Title: Adoptive Cell Therapy for B-Cell Cancers in Patients After Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 070064; 07-C-0064; NCT00445666 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-04-24

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Adoptive Immunotherapy; Tumor Infiltrating Lymphocytes; Refractory Tumor; Resection; B-Cell Malignancies; Chronic Lymphocytic Leukemia; BCL; B-Cell Lymphoid Malignancy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms

INTERVENTIONS:
Drug: Allogeneic Cell Therapy w/ Tumor-derived Lypho

SUMMARY:
Background:

* After allogeneic (donor) stem cell transplantation, a new immune system grows in the patient from the transplanted donor stem cells and lymphocytes (type of immune cell). Donor lymphocytes, unlike the patient s own lymphocytes, often can recognize the patient s tumor cells as being foreign and destroy them.
* It is thought that tumor shrinkage after stem cell transplantation is the result of donor T lymphocytes, or T cells. Some studies show that patients with tumors that have T cells are better able to keep tumor growth in check.
* Patients who have had donor stem cell transplantation may have donor T cells in their tumors that can recognize and fight their cancer. Compared with donor T cells taken directly from the donor and infused into the patient, donor T cells found in patients tumors may be specific for the cancer cells and thus better able to attack tumor. Also, because the T cells found their way to the tumor, they may be less likely to recognize and attack non-tumor tissues than the T cells given in donor lymphocyte infusions.
* The T cells may be especially effective at controlling tumor if they are given an additional stimulus to become active. Costimulation is the name of the body s natural process for providing an extra stimulus, and can be performed on cells in the laboratory. Costimulation can produce large numbers of activated cells that may be able to attack cancer cells and shrink tumors.

Objectives:

-To evaluate the ability of lymphocytes found in tumors from patients who have received donor stem cell transplants to control their tumor growth.

Eligibility:

-Patients between 18 and 75 years of age with a B-cell cancer that has continued to grow or recurred after remission following allogeneic stem cell transplantation. This includes patients who have received transplants from unrelated donors and cord blood.

Design:

* Immune cells are collected from patients blood and blood from their stem cell donor.
* Patients undergo surgery to remove their tumor and a small piece of skin. In the laboratory, donor T cells are isolated from the tumor and costimulated to expand the number of cells and activate them.
* The expanded, activated T cells as infused into the patient.
* Patients have a needle biopsy and possibly surgery to remove a sample of remaining tumor for research studies.
* Patients are followed at the NIH clinic 48 hours after the cell infusion, and again at 1, 2, 4, 8 and 12 weeks after the infusion. Tumor size is monitored every month with CT scans, and possibly also with a PET or bone marrow aspiration and biopsy, for the first 3 months after the cells are infused. Thereafter, visits are less frequent (every 3 months, then every 6 months, and then yearly) during a minimum 5-year follow-up.

DETAILED DESCRIPTION:
Background:

* The prognosis for patients with B-cell lymphoid malignancies (BCL) with relapse or refractory disease after allogeneic hematopoietic stem cell transplantation (AlloHSCT) is poor. Effective therapy for patients who fail withdrawal of immune suppression and administration of donor lymphocyte infusions (DLI) has not been identified.
* In the setting of recurrent or refractory BCL, the immunologic graft-versus-tumor (GVT) effect generated by unmanipulated donor lymphocytes is often not durable and can be accompanied by graft-versus-host disease (GVHD).
* We have hypothesized that lymphocytes found in tumor after alloHSCT are of donor origin, and because they are tumor-derived, they may be tumor-specific in their homing and antigen specificity characteristics. Similarly, inpatients with bone marrow involvement with tumor, the marrow may be enriched with similarly tumor-specific T cells. Further, activation and expansion of these cells through CD3/CD28 costimulation may yield a more effective form of cell therapy than DLI after alloHSCT, with enhanced GVT effects and less GVHD.

Objectives:

* To evaluate the feasibility of isolating and expanding clinically relevant numbers of TDL from patients after alloHSCT.
* To determine the safety, vis-a-vis infusion toxicities and/or GVHD, of administering TDL.

Eligibility:

* Adults with B cell malignancies with tumor that has not responded to successful T cell engraftment after alloHSCT, withdrawal of immune suppression and administration of donor lymphocyte infusion will be eligible for this trial.
* Subjects must have a minimum of 1.5 cm of accessible tumor which is amenable to resection with minimal surgical morbidity and/or bone marrow tumor involvement.

Design:

* Subjects will have accessible lesion surgically resected and/or harvested via bone marrow aspiration.
* Lymphocytes will be liberated and expanded using a co-stimulatory approach with anti-CD3/CD28 magnetic beads to generate TDL and/or marrow-TDL.
* 1.0 x 10(6) - 1.0 x 10(8) TDL will be administered.
* Subjects will be monitored for the development of infusion reactions (in-hospital for 24 hours after infusion), GVHD (weekly for four weeks then monthly) and tumor responses (monthly).
* Two cohorts will be enrolled, with an arm evaluating TDL from resected tumor and an arm to evaluate marrow-TDL from tumor-involved bone marrow. For the TDL arm, 15 to 18 patients and up to 18 donors will be enrolled; for the marrow-TDL arem, 15 patients and up to 15 donors will be enrolled. Both arms will test the primary endpoints of feasibility (with at least 11 of 15 tumors yielding 1.0 x 10(6) TDL/kg meeting defined release criteria) and safety (primarily defined as having a no greater risk of developing grade II-IV acute GVHD by day 28 as standard therapy with unmanipulated DLI).

ELIGIBILITY:
* INCLUSION CRITERIA:

Recipient

1. Patients must have received allogeneic HSCT for B-cell malignancies (BCL), specifically Hodgkin s and non-Hodgkin s lymphomas, chronic lymphocytic leukemias, non T-cell acute lymphoblastic leukemia (B-cell ALL), or multiple myeloma, and must have persistent disease that has failed to respond after a minimum of four weeks to:
2. Donor Engraftment Status: Patients must have had evidence of stable or increasing donor engraftment over the preceding three months and at least 50% donor chimerism in the bone marrow, whole blood and/or circulating CD3+ lymphoid pool.
3. A trial of withdrawal of immunosuppressive therapy, including trials that are discontinued due to development of GVHD
4. Receiving at least one DLI with a minimum T cell dose of 1 x 10(7) CD3+ cells/kg.

   * Patients who have persistent cancer after treatment with an alternative donor alloHSCT (e.g., haploidentical, matched unrelated, umbilical cord blood) or any patient for whom a donor cell product is unavailable and/or timely donor collection is not feasible may be included without failing DLI.
   * Presence of bone marrow involvement with tumor and/or at least one resectable lymph node or other tumor focus that is a minimum of 1.5 cm(3) (estimated size from which at least 1.0 x 106 TNC/kg can be generated):
5. Resectable defined on a case-by-case basis, in collaboration with the Surgical Consult Service.
6. For surgical tumor resection, the expected procedure must be associated with minimal morbidity and minimal hospitalization.
7. In addition to a resectable lesion, there must be at least one other site of disease that permits monitoring for response to therapy.
8. Patients must be 18 75 years of age.
9. ECOG performance status less than or equal to 2 (Karnofsky performance status greater than or equal to 60%).
10. Life expectancy > 3 months.
11. Minimal to no clinical evidence (Grade 0 to 1) of acute GVHD or limited-stage chronic GVHD while off of systemic immunosuppressive therapy for at least four weeks. Subjects who require continued prophylaxis with steroid-sparing agents, e.g.,cyclosporine, or whose disease is controlled with local therapy, e.g., topical steroids or budesonide, will be eligible for enrollment.
12. Provision for a Durable Power of Attorney.
13. Ability to give informed consent.

1.4 Eligibility of Recipients is not contingent upon enrollment of the donor.

Donor

Note: Donor enrollment is not required to meet the primary objectives of this protocol and will not affect eligibility of recipients.

1. Donor must be the same individual whose cells were used as the source for the patient s original stem cell transplant
2. Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis.
3. Donors must be HIV negative, hepatitis B surface antigen negative, and hepatitis C antibody negative.

EXCLUSION CRITERIA:

Recipients

1. Active infection that is not responding to antimicrobial therapy.
2. Active psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent (as determined by Principal Investigator and/or his designee).
3. Pregnant or lactating. Patients of childbearing potential must use an effective method of contraception. The effects of the immunosuppressive medications that could be required to treat GHVD are likely to be harmful to a fetus. The effects upon breast milk are also unknown and may be harmful to an infant.
4. Serum total bilirubin > 2.5 mg/dl, serum ALT and AST values greater than or equal to 2.5 times the upper limit of normal. If the abnormal liver function is attributable to liver involvement by malignancy, patients may be eligible with serum total bilirubin up to 5.0 mg/dl, and serum ALT and AST values up to 5.0 times the upper limit of normal, provided the patient has no evidence of impending hepatic failure (encephalopathy or prothombin time >2 time the upper limit of normal).
5. Minimum absolute neutrophil count of 500 cells/microl, unless attributable to tumor.
6. Untreated leptomeningeal involvement with malignancy.

Donors:

1. History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.
2. History of hypertension that is not controlled by medication, stroke, or severe heart disease (donors with symptomatic angina will be excluded). Donors with a history of coronary artery bypass grafting or angioplasty who are symptom free will receive a cardiology evaluation and be considered on a case-by-case basis.
3. Donors must not be pregnant. Donors of childbearing potential must use an effective method of contraception.
4. Anemia (Hb < 11 gm/dl) or thrombocytopenia (platelets < 100,000 per microl). However, potential donors with Hb levels < 11 gm/dl that is due to iron deficiency will be eligible as long as the donor is initiated on iron replacement therapy. The NIH Clinical Center, Department of Transfusion Medicine will determine the appropriateness of individuals as donors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-01-11; Primary Completion 2013-04-24 (Actual); Study Completion 2013-04-24 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of administering ex-vivo costimulated/expanded tumor-derived lymphocytes (TDL) in patients with persistent or recurrent B-cell lymphoid malignancies (BCL) following treatment with allogeneic hematopoietic stem cell tr...

SECONDARY OUTCOMES:
To determine the safety of administering TDL in patients with persistent/recurrent BCL following alloHSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Hardy, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sahin U, Tureci O, Schmitt H, Cochlovius B, Johannes T, Schmits R, Stenner F, Luo G, Schobert I, Pfreundschuh M. Human neoplasms elicit multiple specific immune responses in the autologous host. Proc Natl Acad Sci U S A. 1995 Dec 5;92(25):11810-3. doi: 10.1073/pnas.92.25.11810. PMID 8524854
- [Background] Russell NH, Byrne JL, Faulkner RD, Gilyead M, Das-Gupta EP, Haynes AP. Donor lymphocyte infusions can result in sustained remissions in patients with residual or relapsed lymphoid malignancy following allogeneic haemopoietic stem cell transplantation. Bone Marrow Transplant. 2005 Sep;36(5):437-41. doi: 10.1038/sj.bmt.1705074. PMID 15980879
- [Background] Fisher RI, Gaynor ER, Dahlberg S, Oken MM, Grogan TM, Mize EM, Glick JH, Coltman CA Jr, Miller TP. Comparison of a standard regimen (CHOP) with three intensive chemotherapy regimens for advanced non-Hodgkin's lymphoma. N Engl J Med. 1993 Apr 8;328(14):1002-6. doi: 10.1056/NEJM199304083281404. PMID 7680764
- [Derived] Hardy NM, Fellowes V, Rose JJ, Odom J, Pittaluga S, Steinberg SM, Blacklock-Schuver B, Avila DN, Memon S, Kurlander RJ, Khuu HM, Stetler-Stevenson M, Mena E, Dwyer AJ, Levine BL, June CH, Reshef R, Vonderheide RH, Gress RE, Fowler DH, Hakim FT, Bishop MR. Costimulated tumor-infiltrating lymphocytes are a feasible and safe alternative donor cell therapy for relapse after allogeneic stem cell transplantation. Blood. 2012 Mar 22;119(12):2956-9. doi: 10.1182/blood-2011-09-378398. Epub 2012 Jan 30. PMID 22289893